CLINICAL TRIAL: NCT02335385
Title: Single Incision Transumbilical Laparoscopic Varicocelectomy: Comparison With the Conventional Laparoscopic Approach.
Brief Title: Single Incision Laparoscopic Varicocelectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Tamer Youssef Mohamed, assistant professor of surgery, Mansoura University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MFM200912
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Varicocele
MeSH Terms: conditions — Varicocele

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SIL-V (Active Comparator): single incision laparoscopic varicocelectomy
  Interventions: Procedure: single incision laparoscopic varicocelectomy
- CTL-V (Active Comparator): conventional transperitoneal laparoscopic varicocelectomy
  Interventions: Procedure: conventional transperitoneal laparoscopic varicocelectomy

INTERVENTIONS:
Procedure: single incision laparoscopic varicocelectomy — bilateral and unilateral varicocelectomy was performed through a single transumbilical flexible SILS port.
  Arms: SIL-V
Procedure: conventional transperitoneal laparoscopic varicocelectomy — bilateral and unilateral varicocelectomy was performed through a conventional 3-ports transperitoneal varicoceletomy
  Arms: CTL-V

SUMMARY:
Conventional laparoscopic varicocelectomy using 3 ports has been used for treatment of varicocele in our department since the nineties. However, the relatively several trocar wounds represent a big challenge against its acceptance by many of our patients who prefer the open approach with one or at least two wounds.

Single incision laparoscopic surgery (SILS), since its introduction in 2007, has been proven to be feasible and effective, with high patient satisfaction rates regarding improved cosmotic outcomes, reduced postoperative pain, and rapid return to normal activities. (10, 11) SILS for varicocelectomy has been reported to be safe and effective alternative to conventional laparoscopic varicocelectomy in a few studies.

ELIGIBILITY:
Inclusion Criteria:

* patients with palpable varicoceles

Exclusion Criteria:

* unfit for anesthesia or laparoscopy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
number of patients with improvement in semen parameters and resolution of testicular pain | 2 years

SECONDARY OUTCOMES:
number of patients developing postoperative complications | 2 years

REFERENCES:
- [Derived] Youssef T, Abdalla E. Single incision transumbilical laparoscopic varicocelectomy versus the conventional laparoscopic technique: A randomized clinical study. Int J Surg. 2015 Jun;18:178-83. doi: 10.1016/j.ijsu.2015.04.048. Epub 2015 May 1. PMID 25937155